CLINICAL TRIAL: NCT00655668
Title: A Phase II, Multicenter, Single-Arm, Open-Label Study to Evaluate the Safety and Efficacy of Single-Agent Lenalidomide (Revlimid®) in Subjects With Relapsed or Refractory T-Cell Non-Hodgkin's Lymphoma
Brief Title: A Phase II Study of Single-Agent Lenalidomide in Subjects With Relapsed Or Refractory T-Cell Non-Hodgkin's Lymphoma
Acronym: EXPECT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision not to pursue as single agent in the study population.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-TCL-001; 2007-002171-13 (EudraCT Number)
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2012-01-05 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: T-cell Non-Hodgkin's Lymphoma
Keywords: NHL, Non-Hodgkin's Lymphoma, T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, Non-Hodgkin | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Open-label, oral lenalidomide monotherapy
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide capsules, 25 mg daily for 21 days in each 28 day cycle
  Other Names: Revlimid

SUMMARY:
This is a Phase II, multicenter, single-arm, open-label study of oral lenalidomide monotherapy administered to subjects with relapsed or refractory T-cell lymphoma. This study will be conducted in two phases: a Treatment Phase and a Follow-up Phase.

Subjects who qualify for enrollment into the study will enter the Treatment Phase and receive single-agent lenalidomide 25 mg once daily on Days 1-21 every 28 days (28-day cycles). Subjects may continue participation in the Treatment Phase of the study for a maximum duration of 24 months, or until disease progression or unacceptable adverse events develop.

All subjects who discontinue the Treatment Phase for any reason will continue to be followed until progression of disease or until next lymphoma treatment is given, whichever comes first, during the Follow-up Phase.

Objectives:

Primary:

• To determine the efficacy of lenalidomide monotherapy in relapsed or refractory T-cell Non-Hodgkin's Lymphoma (NHL). Efficacy will be assessed by measuring the response rate, tumor control rate, duration of response, time to progression and progression free survival.

Secondary:

• To evaluate the safety of lenalidomide monotherapy as treatment for subjects with relapsed or refractory T-cell NHL.

DETAILED DESCRIPTION:
Study was terminated. Study data assessment revealed that study drug is active, but is not likely to be sufficiently active as a single agent in this population for registration purposes.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form.
* Must be ≥ 18 years of age at the time of signing the informed consent form.
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Biopsy-proven T-cell Non-Hodgkin's Lymphoma, either:

  * Peripheral T-cell Lymphoma (PTCL) whatever the subtype, or
  * Cutaneous T-cell Lymphoma (CTCL), but only the subtype mycosis fungoides.
* Relapsed or refractory to previous therapy for T-cell Non-Hodgkin's Lymphoma.
* Must have received at least one prior combination chemotherapy regimen. There is no limit on the number of prior therapies.

Exclusion Criteria:

* Cutaneous T-cell Lymphoma of subtype Sézary Syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2010-03-01 (Actual); Study Completion 2010-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Takeshita, MD, Study Director — Celgene Corporation
Locations (45):
- United States (4):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Cancer Center of Kansas, Wichita, Kansas
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
- Australia (13):
  - The Canberra Hospital Building 3, L 2, Garran, Australian Capital Territory
  - Cancer Therapy Centre, Liverpool, New South Wales
  - Clinical Research Unit Cairns Base Hospital, Cairns, Queensland
  - The Townsville Hospital, Douglas, Queensland
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Ashford Cancer Centre, Ashford, South Australia
  - Royal Adelaide Hospital L3 East Wing, North Terrace, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, 4th Floor, Clive Ward Centre, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - St Vincents Hospital, Fitzroy, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (5):
  - Institute Jules Bordet, Brussels
  - Cliniques Universitaires St Luc, Brussels
  - KUL, Leuven
  - Clinique St Pierre, Ottignies
  - Cliniques universitaires UCL de Mont-Godinne, Yvoir
- France (23):
  - CHU Hôtel Dieu, Nantes, Cedex 01
  - Hôpital Bretonneau, Tours, Cédex 1
  - CHU Hôpital Hôtel Dieu, Angers, Cédex 9
  - Hôpital Claude Huriez, Place de Verdun Cedex, Lille
  - Hôpital Lapeyronie, Cedex, Montpellier
  - Centre Hospitalier Lyon Sud, Lyon Sud, Pierre-Bénite
  - CHRU Hôpitaux de Brabois - Hématologie, Vandœuvre-lès-Nancy, Rue Morvan Cedex
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hôtel Dieu Pavillon Villemur Pasteur, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - Hopital Michallon, Grenoble
  - CHD Les Oudairies, La Roche-sur-Yon
  - CHU Dupuytren, Limoges
  - Hôpital N.D.de Bon Secours, Metz
  - Hôpital Saint-Louis, Paris
  - Hôpital Necker, Paris
  - Hôpital de la Pitié Salpétriere, Paris
  - CHU Rennes Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre René Huguenin, Saint-Cloud
  - Hôpital Purpan, Toulouse
  - Centre Hospitalier, Valence

REFERENCES:
- [Result] Morschhauser F, Fitoussi O, Haioun C, Thieblemont C, Quach H, Delarue R, Glaisner S, Gabarre J, Bosly A, Lister J, Li J, Coiffier B. A phase 2, multicentre, single-arm, open-label study to evaluate the safety and efficacy of single-agent lenalidomide (Revlimid) in subjects with relapsed or refractory peripheral T-cell non-Hodgkin lymphoma: the EXPECT trial. Eur J Cancer. 2013 Sep;49(13):2869-76. doi: 10.1016/j.ejca.2013.04.029. Epub 2013 May 31. PMID 23731832

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruiting began March 2008; first participant enrolled 16 June 2008 and last participant enrolled 29 January 2010.
Pre-assignment Details: Participants with relapsed or refractory, biopsy-proven, T-cell Non-Hodgkin's Lymphoma. Must have received at least one prior chemotherapy regimen which contained two cytotoxic agents.
Groups:
- Single Agent Lenalidomide: Oral lenalidomide 25 mg daily for 21 days every 28 days as tolerated for up to 24 months, until disease progression, or an unacceptable adverse event occurs.
Period: Overall Study
Arm/Group | Single Agent Lenalidomide
Started | 54 (Planned enrollment: 80 participants)
Completed | 0 (Participants dosed up to 24 months, disease progression or unacceptable adverse events developed.)
Not Completed | 54
Not completed — Adverse Event | 6
Not completed — Death | 5
Not completed — Disease Progression | 27
Not completed — Study Terminated | 9
Not completed — Other | 1
Not completed — New Lymphoma Treatment Started | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Agent Lenalidomide
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (11.25)
Age, Customized [Number; unit: participants]
  <=18 years | 0
  >18 years and < = 65 years | 28
  >65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 36
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian/Pacific Islander | 3
  Black | 4
  Hispanic | 1
  White | 45
  Other | 1
  Missing | 0
Region of Enrollment [Number; unit: participants]
  France | 40
  United States | 3
  Belgium | 3
  Australia | 8
Non-Hodgkin's Lymphoma Diagnosis/Histopathology [Number; unit: Participants] — Non-Hodgkin's Lymphoma Diagnosis/Histopathology as assessed by local laboratory at study baseline.
  Cutaneous T-cell lymphoma,mycosis fungoides varient Extranodal Natural Killer (NK)T-cell lymphoma, nasal type Peripheral T-cell lymphoma, not otherwise characterized
  Participants
    Anaplastic large cell lymphoma, primary cutaneous | 1
    Anaplastic large cell lymphoma, primary systemic | 3
    Angioimmunoblastic T-cell lymphoma | 26
    Cutaneous T-cell lymphoma, mycosis fungoides var. | 3
    Extranodal NK T-cell lymphoma, nasal type | 1
    Peripheral T-cell lymphoma, not otherwise charac | 20

OUTCOME MEASURES:

1. Primary Outcome: Participants Categorized by Best Response as Determined by Investigator
Description: Participant response assessed by investigator; criteria by B. Cheson in Journal of Clinical Oncology, 1999 (see article for more detail):
  * Complete Response(CR): Complete disappearance of all detectable disease
  * Complete Response Unconfirmed(CRu): CR, but indeterminate bone marrow
  * Partial Response(PR): >50% decrease in six largest nodes/nodal masses
  * Stable Disease(SD): Less than PR, but not progressive disease
  * Relapsed Disease: In CR/CRu Patients, new lesions seen or increased by >=50% in previous sites
  * Progressive Disease(PD): >=50% increase from low in PR/Non-Responders
Time Frame: Up to 24 months
Population: Intent-to-treat (ITT) Population
Measure: Number; unit: Participants
Arm/Group | Single Agent Lenalidomide
Number analyzed (Participants) | 54
Participants
  Complete Response (CR) | 4
  Complete Response Unconfirmed (CRu) | 2
  Partial Response (PR) | 6
  Stable Disease (SD) | 16
  Progressive Disease (PD) | 16
  No Response Assessment | 9
  Other | 1
  Tumor Control (CR+CRu+PR+SD) | 28

2. Secondary Outcome: Duration of Response
Description: Kaplan-Meier Estimate of duration of response calculated as the time from first computed tomography (CT) Scan or magnetic resonance imaging (MRI) that demonstrates at least a partial response to the first documentation of disease progression, including death due to Non-Hodgkin's Lymphoma.
Time Frame: Up to 24 months
Population: Intent-to-treat (ITT) Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Agent Lenalidomide
Number analyzed (Participants) | 54
Months | 3.55 [3.1562 to 7.6274]

3. Secondary Outcome: Time-to-Progression
Description: Kaplan-Meier estimate of time-to-progression is calculated as the time from the start of study drug therapy to the first documentation of progressive disease.
Time Frame: Up to 24 months
Population: Due to early termination of study, data not analyzed. See outcome #4 for progression-free survival.
Arm/Group | Single Agent Lenalidomide
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-Free Survival
Description: Kaplan-Meier estimate of progression-free survival is defined as the start of study drug therapy to the first observation of disease progression or death due to any cause.
Time Frame: Up to 24 months
Population: Intent-to-treat (ITT) Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Agent Lenalidomide
Number analyzed (Participants) | 54
Months | 2.53 [1.7753 to 4.6356]

5. Secondary Outcome: Safety
Description: Summary of Treatment-Emergent Events in Safety Population (participants with at least one dose of study drug). Events assessed using National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI CTCAE, Version 3: Following is the scale: Grade 1=Mild Adverse Event (AE), Grade 2=Moderate AE, Grade 3=Severe and Undesirable AE, Grade 4=Life-threatening or Disabling AE, and Grade 5=Death Related to AE.)
Time Frame: Up to 24 months
Population: Safety Population (received at least one dose of study drug)
Measure: Number; unit: Participants
Arm/Group | Single Agent Lenalidomide
Number analyzed (Participants) | 54
Participants
  At least 1 adverse event (AE) | 53
  At least 1 AE related to drug | 40
  At least 1 NCI CTCAE Grade 3-4 AE | 34
  At least 1 NCI CTCAE Gr 3-4 AE related to drug | 19
  At least 1 serious adverse event (SAE) | 29
  At least 1 SAE related to drug | 16
  At least 1 AE leading to drug withdrawal (WD) | 21
  At least 1 AE leading to drug interruption/WD | 19

ADVERSE EVENTS:
Time Frame: Up to 24 months
Arm/Group | Single Agent Lenalidomide
Serious Adverse Events (participants affected / at risk) | 29/54
Other Adverse Events (participants affected / at risk) | 53/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent Lenalidomide (N=54)
Anaemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymph Node Pain (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Arrhythmia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Aplasia (Congenital, familial and genetic disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Occular Vasculitis (Eye disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
General Physical Health Deterioration (General disorders) | 3
Hyperthermia (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Pyrexia (General disorders) | 2
Bacterial Sepsis (Infections and infestations) | 1
Cytomegalovirus Infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Neutropenic Infection (Infections and infestations) | 1
Neutropenic Sepsis (Infections and infestations) | 1
Oral Candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pneumonia Pneumococcal (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Septic Shock (Infections and infestations) | 1
Prothrombin Level Decreased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Histiocytosis Haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Kaposi's Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Peripheral T-cell Lymphoma Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour Flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (Nervous system disorders) | 1
Carotid Artery Stenosis (Nervous system disorders) | 1
Cerebral Ischaemia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Transient Ischaemic Attack (Nervous system disorders) | 1
Confusional State (Psychiatric disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Drug Eruption (Skin and subcutaneous tissue disorders) | 1
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent Lenalidomide (N=54)
Anaemia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Abdominal Pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 8
Dry Mouth (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 7
Rectal Haemorrhage (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 11
Fatigue (General disorders) | 5
Oedema Peripheral (General disorders) | 8
Pain (General disorders) | 3
Pyrexia (General disorders) | 14
Weight Decreased (Investigations) | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Tumour Flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Headache (Nervous system disorders) | 6
Paraesthesia (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 5
Renal Failure Acute (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4
Night Sweats (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 6
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.